CLINICAL TRIAL: NCT06800742
Title: Body Composition, Resting Energy Expenditure and Physical Activity in Adolescents With Anorexia Nervosa
Brief Title: Body Composition in Adolescents With Anorexia Nervosa
Acronym: COCOMETANNER
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C409
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia; Resting energy expenditure; Hyperactivity
MeSH Terms: conditions — Anorexia Nervosa; Anorexia; Spasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anorexia Nervosa (AN): Female adolescents with Anorexia Nervosa
  Interventions: Other: Collection of anthropometric and biochemical parameters
- Normal weight: Female normal weight adolescents
  Interventions: Other: Collection of anthropometric and biochemical parameters

INTERVENTIONS:
Other: Collection of anthropometric and biochemical parameters — Collection of anthropometric parameters biochemical parameters basal metabolic rate body composition questionnaires

SUMMARY:
Body Mass Index (BMI) is currently the most widely recommended parameter for identifying underweight subjects. Among eating disorder diseases, anorexia nervosa (AN) is the one with the highest mortality rate and with relapses between 12 and 27%. To date, recovery programs allow approximately 40% of subjects to achieve recovery, 30% demonstrate improvements, and 20% remain chronically affected. These data demonstrate the importance of continuously monitoring changes in weight and body composition of these subjects. Bioelectrical impedance (BIA) is widely used to determine body composition in AN. BIA provides various parameters, such as lean mass (LM), fat mass (FM), total body water (TBW), and phase angle (PhA). Among these parameters, in addition to LM and FM, PhA has also been used to characterize underweight subjects with AN. In addition to the observed relationship between PhA and body composition in individuals with AN, PhA has also been related to the basal metabolic rate (BMR). BMR undergoes changes mainly due to loss of muscle mass and a significant reduction in BMR has been observed in AN subjects. Finally, physical activity represents a significant determinant of body composition and can help regulate BMR.

Therefore, monitoring changes in body composition (LM, FM, and PhA) and indirect indices (lean mass index and fat mass index) using BIA, together with monitoring changes in BMR and physical activity level, could provide important support for the continuous control and definition of the clinical stage of the disease in patients with AN.

The aim of this study is to determine body composition, basal metabolic rate, and level of physical activity in Anorexia Nervosa and normal weight subjects to identify the most consistent parameters to define the clinical stage of the disease in subjects with AN.

DETAILED DESCRIPTION:
Body Mass Index (BMI) is currently the most widely recommended parameter for identifying underweight subjects. Among eating disorder diseases, anorexia nervosa (AN) is the one with the highest mortality rate and with relapses between 12 and 27%. To date, recovery programs allow approximately 40% of subjects to achieve recovery, 30% demonstrate improvements, and 20% remain chronically affected. These data demonstrate the importance of continuously monitoring changes in weight and body composition of these subjects. Bioelectrical impedance (BIA) is widely used to determine body composition in AN. BIA provides various parameters, such as lean mass (LM), fat mass (FM), total body water (TBW), and phase angle (PhA). Among these parameters, in addition to LM and FM, PhA has also been used to characterize underweight subjects with AN. In addition to the observed relationship between PhA and body composition in individuals with AN, PhA has also been related to the basal metabolic rate (BMR). BMR undergoes changes mainly due to loss of muscle mass and a significant reduction in BMR has been observed in AN subjects. Finally, physical activity represents a significant determinant of body composition and can help regulate BMR.

Therefore, monitoring changes in body composition (LM, FM, and PhA) and indirect indices (lean mass index and fat mass index) using BIA, together with monitoring changes in BMR and physical activity level, could provide important support for the continuous control and definition of the clinical stage of the disease in patients with AN.

The aim of this study is to determine body composition, basal metabolic rate, and level of physical activity in Anorexia Nervosa and normal weight subjects to identify the most consistent parameters to define the clinical stage of the disease in subjects with AN.

ELIGIBILITY:
Adolescents with Anorexia Nervosa:

Inclusion Criteria:

* Female sex
* Age range: 12-18 years
* Anorexia nervosa
* Hospitalized at the Division of Auxologia, San Giuseppe Hospital, Istituto Auxologico Italiano, IRCCS, Piancavallo, Italy

Exclusion Criteria:

* Absence of signed informed consent

Adolescents with normal weight:

Inclusion Criteria:

* Female sex
* Age range: 12-18 years
* Normal weight

Exclusion Criteria:

* Absence of signed informed consent

Ages: 12 Years to 18 Years | Sex: Female
Age Groups: Child, Adult
Study Population: 30 female adolescents with Anorexia nervosa, according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), hospitalized at the Division of Auxologia, San Giuseppe Hospital, Istituto Auxologico Italiano, IRCCS, Piancavallo, Italy
  30 normal weight adolescents recruited at the Mountain Sports Study Center of the Department of Medicine, University of Udine, Italy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Fat-free mass | Baseline
  Fat-free mass as assessed by bioelectrical impedance
Fat mass | Baseline
  Fat mass as assessed by bioelectrical impedance
Basal Metabolic Rate | Baseline
  Basal Metabolic Rate as calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy